CLINICAL TRIAL: NCT02304380
Title: Improving Care Coordination for Children With Disabilities Through an Accountable Care Organization
Brief Title: Care Coordination for Children With Disabilities
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 14-2045
Record Dates: First submitted 2014-11-18; First posted 2014-12-01 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2017-10

CONDITIONS: Experiences With Health Care Coordination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The proposed study uses a recent policy change in Ohio as a natural experiment to assess outcomes and experiences of children who qualify for Medicaid under the Aged, Blind, Disabled category and their caregivers in an ACO model of care compared to their previous outcomes and experiences in a traditional fee-for-service model.

DETAILED DESCRIPTION:
Children with disabilities have complex healthcare needs requiring multiple providers in multiple locations. The lack of coordinated care for this vulnerable population leads to poorer outcomes, higher costs, and increased stress and time demands for patients and their caregivers. Traditionally, under arrangements known as fee-for-service, there have been no financial incentives for providers to coordinate care; however, the Affordable Care Act is changing that. Accountable care organizations (ACOs) are groups of healthcare providers that organize in new ways to take responsibility for the care of a defined population. ACOs share in any savings associated with improved quality and efficiency of the care they provide. Although most ACOs currently do not cover children with disabilities, many are considering adding these to the populations they serve. Yet little is known about effectiveness of the care coordination strategies they employ on children with disabilities.

The goal of this research is to assess care coordination for and patient-centered outcomes of children with disabilities (who qualify for Medicaid under the Aged, Blind, Disabled category (ABD) under an ACO as compared with traditional fee-for-service plans. The investigators will use a recent policy change in Ohio that mandates children with disabilities move from traditional fee-for-service Medicaid plans into managed care arrangements such as ACOs. This mandate resulted in 8,000 disabled children automatically becoming part of the nation's largest pediatric ACO.

The investigators will use multiple methods, including focus groups, interviews, a survey, medical record data, and Medicaid claims, to compare patient experiences and care under the ACO with experiences and care under the previous fee-for-service model. What impact will this research have? Our research will inform ACOs about the relative benefits and challenges of coordinating care and improving the health outcomes of children with disabilities and will help those organizations determine whether or not they can adequately serve the needs of this population. In addition, the findings will provide patients and caregivers with valuable information that can help them make decisions when faced with an increasingly common scenario, for example: "The parents of a child with cerebral palsy receive a letter from their state Medicaid program that children are being enrolled in an 'accountable care organization.' How certain can they be that their child's care will be improved? What are the problems that might occur?" The investigators will engage patients, their caregivers, and health system stakeholders throughout the research process. Patient advocates have been involved in the design of our study. A patient advisory panel comprised of caregivers and advocates of disabled children will guide our project by providing advice at quarterly meetings. In addition, the investigators plan to collect data from more than 2,800 patient voices through direct study participation.

ELIGIBILITY:
Inclusion Criteria:

Stakeholder Interviews

- Be associated with the ACO as ACO leadership, a care coordinator, a payor or policy-maker.

Caregiver Interviews

* Currently live in south-central Ohio
* Have lived in south-central Ohio since July 2012
* Be a caregiver of a child ages 3-18 who qualifies for Medicaid under the Aged, Blind, and Disabled category

Focus Groups, Caregivers and Youth

* Currently live in south-central Ohio
* Have lived in south-central Ohio since July 2012
* Be a caregiver of a child ages 3-18 who qualifies for Medicaid under the Aged, Blind, and Disabled (ABD) category, who receives care at Nationwide Children's Hospital, Partners for Kids
* For youth focus groups, be a child ages 14-18 who qualifies for Medicaid under the Aged, Blind, and Disabled category, who is intellectually capable of participating in focus groups, and who receives care at Nationwide Children's Hospital, Partners for Kids

Exclusion Criteria:

* Non-English-speaking
* For youth focus groups, intellectual disabilities that preclude being able to participate in a focus group

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children who qualify for Medicaid under the Aged, Blind, and Disabled category, and their caregivers, who are part of the Nationwide Children's Hospital Partners for Kids Accountable Care Organization (ACO) in Columbus, Ohio.
Sampling Method: Non-Probability Sample
Enrollment: 2188 (Actual)
Dates: Start 2015-03; Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Song, PhD, Principal Investigator — UNC Chapel Hill

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hilligoss B, Tanenbaum SJ, Paul MH, Ferrari RM, Song PH. What makes health services usable?: Insights from a qualitative study of caregivers of children with disabilities. Health Care Manage Rev. 2021 Apr-Jun 01;46(2):111-122. doi: 10.1097/HMR.0000000000000249. PMID 33630503
- [Derived] Song PH, White BA, Chisolm DJ, Berney S, Domino ME. The effect of an accountable care organization on dental care for children with disabilities. J Public Health Dent. 2020 Sep;80(3):244-249. doi: 10.1111/jphd.12375. Epub 2020 Jun 9. PMID 32519336
- [Derived] Sheftall AH, Chisolm DJ, Alexy ER, Chavez LJ, Mangione-Smith RM, Ferrari RM, Song PH. Satisfaction With Care Coordination for Families of Children With Disabilities. J Pediatr Health Care. 2019 May-Jun;33(3):255-262. doi: 10.1016/j.pedhc.2018.08.010. Epub 2018 Nov 16. PMID 30449647

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Claims data records for 64,382 participants were analyzed to address Claims Data Analysis (Aim 3).
Pre-assignment Details: 64,382 met eligibility criteria for inclusion in the claims data analysis which was non-human subjects research.
Groups:
- Accountable Care Organization (ACO) Stakeholder Interviews: Stakeholders from the ACO, insurance payers, departments of health, and representatives from other stakeholder organizations who have knowledge of/experience with care coordination for children with disabilities before and after the 2013 policy change. Informants included leaders, staff, clinicians, representatives Medicaid managed care organizations, and representatives from public health organizations.
- Caregiver & Youth Focus Groups: Caregivers of children with disabilities, and youth (i.e. patients) with disabilities.
  To be eligible to participate, the child (as the participant, OR of the caregiver) must:
  1. Have resided continuously in the region served by the ACO, have been continuously enrolled in Medicaid, and have had Medicaid Aged, Blind, or Disable (ABD) status since at least one year before the policy change;
  2. Be no more than 18 years of age at the time of data collection; and
  3. Have been, at the time of the policy change, at least 14 years of age for youth (patient) focus groups, or 2 years of age for caregiver focus groups.
- Caregiver Interviews: Caregivers of children with disabilities. To be eligible to participate, the caregiver's child must: 1. Have resided continuously in the region served by the ACO, have been continuously enrolled in Medicaid, and have had Medicaid Aged, Blind, or Disabled (ABD) status since at least one year before the policy change; 2. Be no more than 18 years of age at the time of data collection; and 3. Have been, at the time of the policy change, at least 2 years of age.
- Caregiver Survey: Caregivers of children with disabilities who are part of the ACO, and fall into one of three categories: 1) children with ABD status with continuous enrollment since July 2013; 2) children with ABD status with 12 month continuous enrollment as of February 2015; and 3) children who were ABD status as of July 2013 who are no longer eligible for ABD but qualify for Medicaid and are still in the ACO.
- Claims Data-ACO Sample: Claims and enrollment data from the Ohio Medicaid program from August 2011-July 2016 (23 months before entering ACO, 30 months post); dataset includes any child who was ABD status at any point during August 2011-June 2016; dataset does not include children without ABD status. These are unique participants. They were not consented or considered "enrolled".
- Claims Data-Control Sample: Claims and enrollment data from the Ohio Medicaid program from August 2011-July 2016 (23 months before entering ACO, 30 months post); dataset includes children with disabilities on Medicaid under ABD who moved from fee-for-service coverage to non-ACO managed care. Excluded children who enrolled in managed care before the policy change and children not in managed care after the policy change. These are unique participants. They were not consented or considered "enrolled".
Period: Pediatric Claims Data Analysis (Aim 3)
Arm/Group | Accountable Care Organization (ACO) Stakeholder Interviews | Caregiver & Youth Focus Groups | Caregiver Interviews | Caregiver Survey | Claims Data-ACO Sample | Claims Data-Control Sample
Started | 0 | 0 | 0 | 0 | 17356 | 47026
Completed | 0 | 0 | 0 | 0 | 17356 (2,096 Caregivers of the 17,356 claims were included in the Caregiver Survey.) | 47026 (Not included in any other portion of the study.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Pediatric Adult Caregiver Survey (Aim 2)
Arm/Group | Accountable Care Organization (ACO) Stakeholder Interviews | Caregiver & Youth Focus Groups | Caregiver Interviews | Caregiver Survey | Claims Data-ACO Sample | Claims Data-Control Sample
Started | 0 | 0 | 0 | 2096 | 0 | 0
Completed | 0 | 0 | 0 | 2062 (68 Caregivers/Patients of the 2,062 surveyed were included in the Interviews and Focus Group .) | 0 | 0
Not Completed | 0 | 0 | 0 | 34 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 34 | 0 | 0
Period: Interviews & Focus Groups (Aim 1)
Arm/Group | Accountable Care Organization (ACO) Stakeholder Interviews | Caregiver & Youth Focus Groups | Caregiver Interviews | Caregiver Survey | Claims Data-ACO Sample | Claims Data-Control Sample
Started | 0 | 35 | 33 | 0 | 0 | 0
Completed | 0 | 35 | 33 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: ACO Stakeholder Interviews (Aim 1)
Arm/Group | Accountable Care Organization (ACO) Stakeholder Interviews | Caregiver & Youth Focus Groups | Caregiver Interviews | Caregiver Survey | Claims Data-ACO Sample | Claims Data-Control Sample
Started | 24 | 0 | 0 | 0 | 0 | 0
Completed | 24 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ACO Stakeholder Interviews: Stakeholders from the ACO, insurance payers, departments of health, and representatives from other stakeholder organizations who have knowledge of/experience with care coordination for children with disabilities before and after the 2013 policy change. Informants included leaders, staff, clinicians, representatives Medicaid managed care organizations, and representatives from public health organizations.
- Total: Total of all reporting groups
Arm/Group | ACO Stakeholder Interviews | Caregiver & Youth Focus Groups | Caregiver Interviews | Caregiver Survey | Claims Data-ACO Sample | Claims Data-Control Sample | Total
Number analyzed (Participants) | 24 | 35 | 33 | 2062 | 17356 | 47026 | 66536
Age, Categorical [Count of Participants; unit: Participants] — Population: Age was missing for 1 person from the focus groups.
  Age was missing for 5 persons from the caregiver survey.
  No data were collected for the ACO stakeholder arm/groups.
  Participants
    number analyzed (Participants) | 0 | 34 | 33 | 2057 | 17356 | 47026 | 66506
    <=18 years |  | 2 | 0 | 0 | 17356 | 47026 | 64384
    Between 18 and 65 years |  | 31 | 33 | 2019 | 0 | 0 | 2083
    >=65 years |  | 1 | 0 | 38 | 0 | 0 | 39
Age, Continuous [Mean (Full Range); unit: years] — Population: Demographic data for ACO Stakeholder Interviews were not collected. Age was missing for 1 person from the focus groups. Age was missing for 5 persons from the caregiver survey.
  years
    number analyzed (Participants) | 0 | 34 | 33 | 0 | 17356 | 47026 | 64449
    (all) |  | 38.6 [17 to 73] | 40 [27 to 64] |  | 12.3 [0 to 18] | 12.7 [0 to 18] | 12.6 [0 to 73]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We collected 2062 caregiver surveys. For the analyses, we dropped one survey because the participant's demographic data on the caregiver survey did not match medical record data. Because we dropped one survey, the final sample size for analysis was 2061. Did not collect demographic data for the ACO stakeholder interview arm/group.
  Participants
    number analyzed (Participants) | 0 | 35 | 33 | 2061 | 17356 | 47026 | 66511
    Female |  | 33 | 32 | 1908 | 5901 | 16224 | 24098
    Male |  | 2 | 1 | 153 | 11455 | 30802 | 42413
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: We did not collect demographic data on our key informants. Ethnicity data are not available for the Claims Data-ACO Sample/Claims Data Control Sample.
  Participants
    number analyzed (Participants) | 0 | 35 | 33 | 2061 | 17356 | 47026 | 66511
    Hispanic or Latino |  | 0 | 0 | 76 | 0 | 0 | 76
    Not Hispanic or Latino |  | 35 | 30 | 1981 | 0 | 0 | 2046
    Unknown or Not Reported |  | 0 | 3 | 4 | 17356 | 47026 | 64389
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: We did not collect demographic data on our key informants.
  Participants
    number analyzed (Participants) | 0 | 35 | 33 | 2061 | 17356 | 47026 | 66511
    American Indian or Alaska Native |  | 0 | 0 | 10 | 29 | 68 | 107
    Asian |  | 0 | 0 | 10 | 141 | 209 | 360
    Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 2 | 4 | 57 | 63
    Black or African American |  | 12 | 13 | 628 | 5102 | 21633 | 27388
    White |  | 23 | 20 | 1265 | 11306 | 23030 | 35644
    More than one race |  | 0 | 0 | 67 | 0 | 0 | 67
    Unknown or Not Reported |  | 0 | 0 | 79 | 774 | 2029 | 2882
Region of Enrollment [Count of Participants; unit: Participants] — Population: We collected 2062 caregiver surveys. For the analyses, we dropped one survey because the participant's demographic data on the caregiver survey did not match medical record data. Because we dropped one survey, the final sample size for analysis was 2061.
  Participants
    United States: number analyzed (Participants) | 24 | 35 | 33 | 2061 | 17356 | 47026 | 66535
    United States | 24 | 35 | 33 | 2061 | 17356 | 47026 | 66535

OUTCOME MEASURES:

1. Primary Outcome: Percent of Caregivers Who Reported That Their Child Has a Designated Care Coordinator
Description: This outcome was measured using the validated tool, "Family Experiences with Coordination of Care" (FECC) survey. The FECC survey is made up of 20 separate and independent quality indicators related to care coordination for children with medical complexity. To be included in the denominator for this measure, caregivers first had to report that their child visited more than one doctor's office or used more than one kind of health care service in the 12 months prior to the survey date. To measure the percent of caregivers who reported that their child has a designated care coordinator among those in the denominator, caregivers needed to have answered yes to one of the following two questions: "Did anyone in the main provider's office help you to manage your child's care or treatment from different doctors or care providers?" or "Did anyone outside of the main provider's office help you to manage your child's care or treatment from different doctors or care providers?".
Time Frame: 12 month lookback from time of survey
Population: To be included in the analysis for this measure, caregivers first had to report that their child visited more than one doctor's office or used more than one kind of health care service in the 12 months prior to the survey date.
Measure: Count of Participants; unit: Participants
Groups:
- Caregiver Survey: Caregivers of children with disabilities who are part of the Accountable Care Organization (ACO), and fall into one of three categories: 1) children with Medicaid Aged, Blind, or Disabled (ABD) status with continuous enrollment since July 2013; 2) children with ABD status with 12 month continuous enrollment as of February 2015; and 3) children who were ABD status as of July 2013 who are no longer eligible for ABD but qualify for Medicaid and are still in the ACO.
Arm/Group | Caregiver Survey
Number analyzed (Participants) | 1201
Participants | 864

2. Secondary Outcome: Percent of Caregivers Who Reported That Their Care Coordinator Asked About Caregiver Concerns and Changes in the Child's Health
Description: This outcome was measured using FECC survey. To be included in the denominator for this measure, caregivers first had to report that their child visited more than one doctor's office or used more than one kind of health care service in the 12 months prior to the survey date AND were contacted by their care coordinator in the past 3 months. Caregivers then had to respond positively to both of the following two questions: "In the last 3 months, when the person who helped you with managing your child's care contacted you, how often did he or she ask if you had any concerns about your child's health or treatment?" and "In the last 3 months, when the person who helped you with managing your child's care contacted you, how often did he or she ask if your child's health had changed in any way?".
Time Frame: 3 month lookback from time of survey
Population: Percentage of participants who reported that their child visited more than one doctor's office or used more than one kind of health care service in the last 12 months and who were contacted by their care coordinator in the past 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver Survey
Number analyzed (Participants) | 435
Participants | 261

3. Secondary Outcome: Percent of Caregivers Who Reported Receiving a Comprehensive Written After-visit Summary in the Past 12 Months
Description: This outcome was measured using FECC survey. To be included in the denominator for this measure, caregivers first had to report that they received a written after-visit summary from their child's main provider's office. Caregivers then had to report that the written after-visit summary contained all of the following elements: current problem list, current medication list, drug allergies, specialists involved in the child's care, planned follow-up, and what to do for problems related to the outpatient visit.
Time Frame: 12 month lookback from time of survey
Population: To be included in the analysis for this measure, caregivers first had to report that they received a written after visit summary in the past 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver Survey
Number analyzed (Participants) | 1259
Participants | 523

4. Secondary Outcome: Percent of Caregivers Who Reported That Their Child's Primary Care Provider Created a Shared Care Plan for Their Child
Description: This outcome was measured using FECC survey. Caregivers needed to have answered yes to the following question: "Has the main provider created a shared care plan for your child?".
Time Frame: 12 month lookback from time of survey
Population: Participants who responded to the question, "Has the main provider created a shared care plan for your child?"
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver Survey
Number analyzed (Participants) | 1983
Participants | 985

5. Secondary Outcome: Use of One or More Well-child Visits <=6 Years Old
Description: Indicator of use of an age-appropriate well-child visit for children less than or equal to 6 years of age according to the Healthcare Effectiveness Data and Information Set (HEDIS) due to the Accountable Care Organization (ACO). ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of visits in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: The overall data included children up to 18 years of age; however, only those children less than or equal to 6 years of age were included in the analysis.
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 4,297 | 11,397
person-year observations | 9,235 | 25,106
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in differences = -0.0064, 95% CI 2-sided [-0.0469 to 0.0340] — Linear model difference in incidences

6. Secondary Outcome: Use of One or More Well-child Visits >=12 Years Old
Description: Use of an age-appropriate well-child visits for children greater than or equal to 12 years of age according to the Healthcare Effectiveness Data and Information Set (HEDIS) due to the ACO. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of visits in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: Patients who are greater than or equal to 12 years of age
Measure: Number; unit: person-year observations
Groups:
- Claims Data-ACO Sample: Claims and enrollment data from the Ohio Medicaid program from August 2011-July 2016 (23 months before entering ACO, 30 months post); dataset includes any child who was ABD status at any point during August 2011-June 2016; dataset does not include children without ABD status
- Claims Data-Control Sample: Claims and enrollment data from the Ohio Medicaid program from August 2011-July 2016 (23 months before entering ACO, 30 months post); dataset includes children with disabilities on Medicaid under ABD who moved from fee-for-service coverage to non-ACO managed care. Excluded children who enrolled in managed care before the policy change and children not in managed care after the policy change.
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 10,236 | 29,350
person-year observations | 24,342 | 72,803
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in Differences = 0.0506, 95% CI 2-sided [0.0290 to 0.0722] — Linear model difference in incidences

7. Secondary Outcome: Indicator of Use of Primary Care
Description: An indicator of one or more outpatient visits to primary care providers (PCP). ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of visits in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: Please note that the number of person-year observations is the same for multiple outcomes - as long as a child is enrolled in Medicaid that year, we would have the same number of observations.
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 17,356 | 47,026
person-year observations | 49,358 | 142,579
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in Differences = -0.0005, 95% CI 2-sided [-0.0109 to 0.0099] — Linear model difference in incidences

8. Secondary Outcome: Use of Outpatient Medicaid Visits to Other Behavioral Health Providers
Description: Use of one or more outpatient visits to other mental health specialists besides psychiatrists. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of visits in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: as for outcome 7
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 17,356 | 47,026
person-year observations | 49,358 | 142,579
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in differences = -0.0207, 95% CI 2-sided [-0.0318 to 0.0096]

9. Secondary Outcome: Emergency Department Use
Description: Indicator of utilization of emergency department. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of visits in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: as for outcome 7
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 17,356 | 47,026
person-year observations | 49,358 | 142,579
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in differences = 0.0163, 95% CI 2-sided [0.0036 to 0.0289] — Linear model difference in incidences

10. Secondary Outcome: Use of Hospitalizations
Description: Indicator of hospitalization for patients. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of visits in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: as for outcome 7
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 17,356 | 47,026
person-year observations | 49,358 | 142,579
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in differences = 0.0046, 95% CI 2-sided [-0.0020 to 0.0111]; Linear model difference in incidences

11. Secondary Outcome: Follow-up Within 7 Days After Hospitalization
Description: Indicator of follow-up within 7 days after hospitalization. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of visits in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 30 months post
Population: Children who were hospitalized
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 3,950 | 11,877
person-year observations | 10,602 | 31,968
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in differences = 0.0151, 95% CI 2-sided [-0.0129 to 0.0431] — Linear model difference in incidences

12. Secondary Outcome: Follow-up Within 30 Days After Hospitalization
Description: Indicator of having follow-up within 30 days after hospitalization. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of visits in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: Children who were hospitalized
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 3,950 | 11,877
person-year observations | 10,602 | 31,968
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in Differences = -0.0066, 95% CI 2-sided [-0.0328 to 0.0197] — Linear model difference in incidences

13. Secondary Outcome: Hospital Readmissions Within 30 Days After Discharge
Description: Indicator of hospital readmissions within 30 days after discharge. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control group include any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of readmissions in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: Children who were hospitalized
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 3,950 | 11,877
person-year observations | 10,602 | 31,968
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in Differences = -0.0105, 95% CI 2-sided [-0.0374 to 0.0163] — Linear model difference in incidences

14. Secondary Outcome: Hospitalization for Mental Illness
Description: Indicator of hospitalization for mental illness for patients. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of visits in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: Children hospitalized for mental illness. Please note that the number of person-year observations is the same for multiple outcomes - as long as a child is enrolled in Medicaid that year, we would have the same number of observations.
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 17,356 | 47,026
person-year observations | 49,358 | 142,579
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in Differences = 0.0006, 95% CI 2-sided [-0.0031 to 0.0044] — Linear model difference in incidences

15. Secondary Outcome: Follow-up Within 7 Days After Hospitalization for Mental Illness
Description: Indicator of follow-up within 7 days after hospitalization for mental illness. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of visits in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: Children hospitalized for mental illness
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 818 | 3,376
person-year observations | 1,484 | 7,409
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Linear model difference in incidences; Difference in Differences = -0.0293, 95% CI 2-sided [-0.1025 to 0.0440]

16. Secondary Outcome: Follow-up Within 30 Days After Hospitalization for Mental Illness
Description: Indicator of follow-up within 30 days after hospitalization for mental illness. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of visits in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: Children who were hospitalized for mental illness
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 818 | 3,376
person-year observations | 1,484 | 7,409
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in Differences = -0.0579, 95% CI 2-sided [-0.1492 to 0.0116] — Linear model difference in incidences

17. Secondary Outcome: Medication Use - Antidepressants
Description: Indicator of antidepressant medication fills. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of medication fills in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: as for outcome 7
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 17,356 | 47,026
person-year observations | 49,358 | 142,579
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in differences = 0.0072, 95% CI 2-sided [0.0010 to 0.0134] — Linear model difference in incidences

18. Secondary Outcome: Medication Use - Anticonvulsants
Description: Indicator of use of anticonvulsant medication fills. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of medication fills in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: as for outcome 7
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 17,356 | 47,026
person-year observations | 49,358 | 142,579
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in Differences = 0.0058, 95% CI 2-sided [0.0009 to 0.0107]

19. Secondary Outcome: Medication Use - Anti-anxiety Medications
Description: Indicator of use of anti-anxiety medication. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of medication fills in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: as for outcome 7
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 17,356 | 47,026
person-year observations | 49,358 | 142,579
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in Differences = 0.0054, 95% CI 2-sided [0.0001 to 0.0106] — Linear model difference in incidences

20. Secondary Outcome: Medication Use - Anti-psychotic Medications
Description: Indicator of use of anti-psychotic medication. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of medication fills in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: as for outcome 7
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 17,356 | 47,026
person-year observations | 49,358 | 142,579
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in Differences = -0.0039, 95% CI 2-sided [-0.0096 to 0.0017] — Linear model difference in incidences

21. Secondary Outcome: Medication Use - ADHD Medications
Description: Indicator of use of attention deficit hyperactivity disorder (ADHD) medications. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of medication fills in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: as for outcome 7
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 17,356 | 47,026
person-year observations | 49,358 | 142,579
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in Differences = -0.0110, 95% CI 2-sided [-0.0178 to -0.0043] — Linear model difference in incidences

22. Secondary Outcome: Medication Use - Asthma Medications
Description: Indicator of asthma medications fills. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of medication fills in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: as for outcome 7
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 17,356 | 47,026
person-year observations | 49,358 | 142,579
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in Differences = 0.0026, 95% CI 2-sided [-0.0036 to 0.0086] — Linear model difference in incidences

23. Secondary Outcome: Follow-up Within 30 Days After ADHD Prescription
Description: Indicator of one or more follow-up visits within 30 days after ADHD (attention deficit hyperactivity disorder) prescription. ACO sample includes any child who was ABD at any point during the study time period enrolled in the ACO. Control sample includes any child who was ABD and who moved from fee-for-service coverage to non-ACO managed care during the study period. Transforms a count of actual number of visits in a year to an indicator that the number was greater than zero.
Time Frame: 23 months before policy change (2013), 36 months post
Population: Children who received ADHD (attention deficit hyperactivity disorder) prescription
Measure: Number; unit: person-year observations
Arm/Group | Claims Data-ACO Sample | Claims Data-Control Sample
Number analyzed (Participants) | 6,605 | 18,163
person-year observations | 75,757 | 214,253
Statistical Analysis 1: Comparison: Claims Data-ACO Sample vs Claims Data-Control Sample; Test type: Other; Difference in differences = 0.0197, 95% CI 2-sided [0.0110 to 0.0284] — Linear model difference in incidences

ADVERSE EVENTS:
Time Frame: 14 months total, from March 2015 (beginning of stakeholder interviews) to May 2016 (all focus groups and interviews completed).
Description: The Claims Data ACO and Claims Data Control sample were not monitored for adverse events.
Arm/Group | Accountable Care Organization (ACO) Stakeholder Interviews | Caregiver & Youth Focus Groups | Caregiver Interviews | Caregiver Survey | Claims Data-ACO Sample | Claims Data-Control Sample
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/35 | 0/33 | 0/2096 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/35 | 0/33 | 0/2096 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/24 | 0/35 | 0/33 | 0/2096 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT02304380/Prot_SAP_000.pdf